CLINICAL TRIAL: NCT00373750
Title: In-home Prevention of SA Risks for Native Teen Families
Brief Title: Cradling Our Future Through Family Strengthening Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Allison Barlow, Assistant Scientist, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DA019042-01A1 (NIH); 1R01DA019042-01A1 (NIH)
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Substance Abuse; Post-partum Depression; Depression
Keywords: Native American health; Teen pregnancy; Family strengthening; Substance abuse prevention; Injury prevention
MeSH Terms: conditions — Substance-Related Disorders; Depression, Postpartum; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Spirit Intervention (Experimental): The Family Spirit Intervention included 43 structured lessons and followed a culturally congruent format. Positive parenting lessons were focused on reducing behaviors (i.e., poor monitoring; coercive interactions;harsh, unresponsive, or rejecting parenting; and abuse/ neglect) associated with early childhood behavior problems, including externalizing, internalizing, and dysregulation problems.
  Interventions: Procedure: Family Spirit Intervention
- Optimized Standard Care Control Group (No Intervention): Optimized standard care consisted of transportation to recommended prenatal and well-baby clinic visits, pamphlets about child care and community resources, and referrals to local services. It also addressed access barriers to health care for young mothers and children, and it overcame concerns that home-visiting programs have operated in parallel, not in partnership, with pediatric care. Family health liaisons conducted the optimized standard care and were not trained in the Family Spirit intervention, to avoid contamination of the control condition.

INTERVENTIONS:
Procedure: Family Spirit Intervention — The Family Spirit Intervention was developed over a decade through community-based participatory research.The intervention content included 43 structured lessons and followed a culturally congruent format.
  Arms: Family Spirit Intervention

SUMMARY:
The purpose of this study is to determine whether an in-home, paraprofessional-delivered family strengthening curriculum entitled Family Spirit is effective at increasing parental competence, improving maternal outcomes and improving childhood outcomes in a sample of at-risk teen mothers living in four Native American reservation communities. The effectiveness of the Family Spirit curriculum will be determined by comparing outcomes of mothers who receive the intervention plus assisted transportation to prenatal and well baby visits (called Optimal Standardized Care) to mothers who receive only Optimal Standardized Care. Outcomes will be assessed at multiple intervals over the course of a 39-month study period.

DETAILED DESCRIPTION:
American Indians (AIs) in reservation communities have the poorest health, education and socioeconomic status of any racial or ethnic group in the U.S., placing AI youth at increased risk for drug abuse (alcohol, marijuana, tobacco, etc.) and adverse health and behavior outcomes. This study focuses on one of the most vulnerable groups of reservation-based AIs-AI teen mothers and their children.

Over the past two decades a number of research-based health promotion and drug abuse prevention programs for youth have been found to be effective. Of these, parenting interventions have been found to be more effective than other types of interventions. Home visiting programs for young, high-risk mothers have been designed to impact a wide range of outcomes--parenting, child and maternal health and behavior outcomes. More than 40 studies have been published since 1982 supporting the short and long-term efficacy of home visiting programs delivered during pregnancy and early childhood for low-income families. Positive outcomes have been demonstrated for improved parenting and the home environment; increased social support for mothers and children from extended family members and improved maternal health and behavior outcomes; increased birth spacing; improved children's health and behavior outcomes; prevention of child abuse and neglect; and reduced drug use.

AI teen mothers and their offspring are arguably the most vulnerable and underserved population at risk for drug abuse and adverse health and behavior outcomes in the U.S. Given their high-risk status, pregnant AI teens are likely to benefit from a parenting-focused, home visiting intervention. Cultural support for developing individual strengths through a family-based model and the noted cultural relevance of employing AI paraprofessionals are expected to enhance participants' outcomes. As nearly half of AI women begin child-bearing in adolescence, improvement in outcomes of teen mothers and their offspring could substantially impact the public health and welfare of AI communities.

Both nurses and paraprofessionals have been utilized in effective home visiting programs. However, the shortage of indigenous nurses in reservation communities renders an AI nurse-delivered, home visiting intervention unfeasible for the participating communities at this time. Further, young AI women's discomfort with health care delivered by non-Indians and the potential for cultural barriers with non-Indian home visitors provides an additional rationale for AI paraprofessionals as home visitors.

Successful home visiting programs maintain a standard for frequency and dosage of visits, employ strategies for participant retention, provide intensive training, frequent direct supervision and intensive quality assurance measures. For this study, we will maintain the highest standards for dosage, retention strategies, home visitor training and supervision, and quality assurance. The core content of the curriculum is based on American Academy of Pediatrics' comprehensive guidelines for preparing mothers to care for infants and young children, with cultural adaptations derived through guidance from our Native Advisory Board and an iterative process of community input.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant AI females aged 12 to 19 years old at time of conception.
* Gestational age of 28 weeks or less (in order to complete intervention prior to delivery).
* Parent/guardian consent for youth under 18 years old.
* Reside within 1-hour transportation range (50 miles) of the local Indian Health Service medical facility.

Exclusion Criteria:

* Current participation in other mental or behavior health research project.
* Factors that preclude full participation, identified at baseline and after caseness review, including: unstable and severe medical, psychiatric or drug use problem; acute suicidal or homicidal ideation requiring immediate intervention; recent, severe stressful life event such as physical or sexual abuse, or victim of a violent crime that requires specific and high intensity intervention or out of home placement; or chronic pattern of unstable caretakers or living situation.

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 322 (Actual)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Increase in parental competence at nine intervals over 39 month study period | birth-3 year postpartum

SECONDARY OUTCOMES:
Differences in social and emotional competence, and internalizing, externalizing and regulatory problems for children between ages 12-36 months | birth-3 year postpartum
Moderators and mediators of intervention response for mothers and children. | birth-3 year postpartum
Increase in maternal outcomes at nine intervals over 39 month study period | birth-3 year postpartum
Improved childhood outcomes at nine intervals over 39 month study period | birth-3 year postpartum

CONTACTS AND LOCATIONS:
Overall Officials: John Walkup, MD, Principal Investigator — Johns Hopkins University; Allison Barlow, MA, MPH, Study Director — Johns Hopkins Center for American Indian Health
Locations (5):
- United States (5):
  - Johns Hopkins Center for American Indian Health, Fort Defiance, Arizona
  - Johns Hopkins Center for American Indian Health, San Carlos, Arizona
  - Johns Hopkins Center for American Indian Health, Tuba City, Arizona
  - Johns Hopkins Center for American Indian Health, Whiteriver, Arizona
  - Johns Hopkins Center for American Indian Health, Baltimore, Maryland

REFERENCES:
- [Background] Barlow A, Varipatis-Baker E, Speakman K, Ginsburg G, Friberg I, Goklish N, Cowboy B, Fields P, Hastings R, Pan W, Reid R, Santosham M, Walkup J. Home-visiting intervention to improve child care among American Indian adolescent mothers: a randomized trial. Arch Pediatr Adolesc Med. 2006 Nov;160(11):1101-7. doi: 10.1001/archpedi.160.11.1101. PMID 17088511
- [Derived] Haroz EE, Ingalls A, Kee C, Goklish N, Neault N, Begay M, Barlow A. Informing Precision Home Visiting: Identifying Meaningful Subgroups of Families Who Benefit Most from Family Spirit. Prev Sci. 2019 Nov;20(8):1244-1254. doi: 10.1007/s11121-019-01039-9. PMID 31432381
- [Derived] Barlow A, Mullany B, Neault N, Goklish N, Billy T, Hastings R, Lorenzo S, Kee C, Lake K, Redmond C, Carter A, Walkup JT. Paraprofessional-delivered home-visiting intervention for American Indian teen mothers and children: 3-year outcomes from a randomized controlled trial. Am J Psychiatry. 2015 Feb 1;172(2):154-62. doi: 10.1176/appi.ajp.2014.14030332. Epub 2014 Oct 31. PMID 25321149
- [Derived] Barlow A, Mullany B, Neault N, Compton S, Carter A, Hastings R, Billy T, Coho-Mescal V, Lorenzo S, Walkup JT. Effect of a paraprofessional home-visiting intervention on American Indian teen mothers' and infants' behavioral risks: a randomized controlled trial. Am J Psychiatry. 2013 Jan;170(1):83-93. doi: 10.1176/appi.ajp.2012.12010121. PMID 23409290